CLINICAL TRIAL: NCT06753253
Title: Effects of Low, Moderate, and High Intensity Exercise on Executive Function, Functional Impairment, and Symptom Severity in ADHD
Brief Title: Effects of Exercise Intensity on ADHD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1265
Record Dates: First submitted 2024-12-05; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Disorder with Hyperactivity; Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Intensity (Experimental): The low intensity arm will perform 20 minutes of steady-state cycling on an airdyne bike. Intensity will be confirmed with continuous heart rate measurement, and heart rate should not exceed 65% of maximal heart rate (220-age) in this arm.
  Interventions: Behavioral: Cycling Exercise
- Moderate Intensity (Experimental): The moderate intensity arm will perform 20 minutes of steady-state cycling on an airdyne bike, maintaining heart rate between 65-85% of maximal heart rate.
  Interventions: Behavioral: Cycling Exercise
- High-Intensity (Experimental): The high-intensity arm will perform a 3-minute steady-state cycling warm up on an airdyne bike, followed by 16 minutes of high intensity interval training (HIIT) cycling. The HIIT protocol consists of alternating periods of 20 seconds of high-intensity effort and 120 seconds of return to low-intensity steady-state cycling. The heart rate goal to ensure high-intensity effort is to maintain heart rate > 85% maximal heart rate during the 20 second high-intensity bursts.
  Interventions: Behavioral: Cycling Exercise

INTERVENTIONS:
Behavioral: Cycling Exercise — Each arm will perform a 20-minute cycling intervention on an airdyne bike at different exercise intensity levels. Participants will perform the intervention three times over the course of one week.

SUMMARY:
This project investigates the effects of a bicycling exercise at three levels of exercise intensity (low, moderate, and high) on attention deficit/hyperactivity disorder (ADHD) in college students. Specifically, the outcomes of interest in this study are self-reported executive functioning, self-reported functional impairment, and ADHD symptom severity. The hypothesis is that exercise will improve executive functioning, while reducing functional impairment and ADHD symptom severity, and that this response will be most pronounced in the high-intensity exercise group.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of attention deficit/hyperactivity disorder (ADHD) Age 18-16 Student at Kent State University

Exclusion Criteria:

seizures/epilepsy syncope asthma chronic obstructive pulmonary disease (COPD) restrictive lung disease adult respiratory distress syndrome (ARDS) heart problems/defects/heart failure/valve problems liver/kidney disease diabetes mellitus current pregnancy

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Self-Reported Executive Function | The BDEFS will be assessed on the first day of participation in an exercise intervention (session 1) and again on the last day of the intervention (session 3). Session 1 occurs on a Monday, session 2 on a Wednesday, and Session 3 on a Friday.
  Self-reported executive function will be measured using a modified version of the Barkley Executive Function Scale (BDEFS)
Self-Reported Functional Impairment | The BFIS will be assessed on the first day of participation in an exercise intervention (session 1) and again on the last day of the intervention (session 3). Session 1 occurs on a Monday, session 2 on a Wednesday, and Session 3 on a Friday.
  Self-Reported Functional Impairment will be measured using a modified version of the Barkley Functional Impairment Scale (BFIS)
Self-Reported ADHD Symptom Severity | The BAARS-IV will be assessed on the first day of participation in an exercise intervention (session 1) and again on the last day of the intervention (session 3). Session 1 occurs on a Monday, session 2 on a Wednesday, and Session 3 on a Friday.
  Self-Reported ADHD Symptom Severity will be measured using the Barkley Adult ADHD Rating Scale IV (BAARS-IV)

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No